CLINICAL TRIAL: NCT06858072
Title: Comparative Effects of Transverse Friction Massage Versus Instrument-assisted Soft Tissue Mobilization on Pain, Range of Motion, and Posture in Patients With Quadratus Lumborum Syndrome
Brief Title: Transverse Friction Massage Versus Instrumented Assisted Soft Tissue Mobilization in Quadratus Lumborum Syndrome
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Riphah International University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: REC/RCR &AHS/24/0127
Record Dates: First submitted 2025-02-20; First posted 2025-03-05 (Actual); Last update posted 2025-03-05 (Actual); Status verified 2025-03

CONDITIONS: Quadratus Lumborum Syndrome

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Instrument assisted soft tissue mobilization (Experimental): IASTM (Instrument-Assisted Soft Tissue Mobilization) in four specific body areas for four weeks. The quadratus lumborum, posterior fascia, sacrum, hip lateral rotators, and hamstring bilaterally
  Interventions: Other: Instrument assissted soft tissue mobilization(IASTM)
- Transverse friction massage (Active Comparator): therapist will perform the transverse friction massage using their thumb to apply pressure across the muscle fibers of Quadratus Lumborum
  Interventions: Other: Transverse friction massage

INTERVENTIONS:
Other: Instrument assissted soft tissue mobilization(IASTM) — IASTM (Instrument-Assisted Soft Tissue Mobilization) in four specific body areas. The quadratus lumborum, posterior fascia, sacrum, hip lateral rotators, and hamstring bilaterally were these areas. The subjects were asked to kneel directly on the bed to stimulate the lumbar posterior muscles erector spinae (iliocostalis, longissimus), lumborum, and multifidus. At the same time, the IASTM treatment was applied to the rear fascia. The same treatment was applied to the sacrum while the subject kneeled on the bed. For hip lateral rotators, the IASTM treatment was applied to the gluteus maximus and gluteus medius while kneeling in a prone position with knee and hip flexion. Similarly, for the hamstring bilaterally, the IASTM treatment was applied to the biceps femoris, semitendinosus, and semimembranosus while in a prone position. The instrument was used for about 20 seconds in a direction parallel to the muscle fibers being treated and then for an additional 20 sec perpendicular to fibres
  Arms: Instrument assisted soft tissue mobilization
Other: Transverse friction massage — patient was lying prone while the therapist administered a transverse friction massage to the affected area. Before the massage, the therapist cleansed and dried the place to be treated, ensuring it was free of dirt or debris. The therapist used their palpation skills to locate the site of pain and apply the massage technique accordingly. The therapist performed the transverse friction massage using their thumb to apply pressure across the muscle fiber, with each repetition lasting for two minutes
  Arms: Transverse friction massage

SUMMARY:
To find effective therapeutic interventions for QLS, a study is being conducted to compare the efficacy of two promising techniques: Transverse Friction Massage (TFM) and Instrument-Assisted Soft Tissue Mobilization (IASTM) . Participants will be randomly assigned to either the TFM or IASTM groups. Outcome measures will be collected before and after the intervention, including pain levels assessed through NPRS, range of motion using inclinometer and posture by measuring leg length discrepancy with tape method.Non probability convenience sampling will be used and 34 partcipants will be randomly allocated in two groups after meeting inclusion criteria.Both groups will receive hotpack for 10-15min.Stretching quadratus lumborum will also be performed with strengthening on the opposite side of affected quadratus lumborum.This methodology provides a solid assessment of the effectiveness of TFM and IASTM for Quadratus Lumborum Syndrome therapy.

ELIGIBILITY:
Inclusion Criteria:

* Age group between 18-40years
* Males only with target population was office workers
* NPRS>4
* Patients with a positional fault of the pelvis (lateral tilt)
* Patients having chronic LBP for more than six months
* Hyperirritable spot or taut band
* Positive jump sign for trigger points/ Referred pain related to the trigger point area
* Positive Lewis's functional palpation test for QL overactivity
* At least one trigger point in Quadratus lumborum
* Leg length discrepancy due to QL tightness

Exclusion Criteria:

* Congenital or acquired spinal deformities
* Spinal stenosis or radiculopathy
* Diagnosed disc prolapse
* Rheumatoid arthritis
* Any malignancy
* Recent history of surgery less than three months
* Acute infections

Ages: 18 Years to 40 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes — Males 18-40years
Enrollment: 34 (Actual)
Dates: Start 2023-05-02 (Actual); Primary Completion 2023-12-23 (Actual); Study Completion 2024-07-02 (Actual)

PRIMARY OUTCOMES:
Numeric Pain rating scale(NPRS) | 8 weeks
  The Numeric Pain Rating Scale (NPRS-11) has been widely used clinically to assess pain. Universal pain screening with a 0-10 pain intensity numeric pain rating scale (NPRS) has been widely implemented in primary care. The current study will use this scale to measure pain in the lumbosacral joint. A numerical pain rating scale (NPRS) requires patients to rate their pain on a defined scale. For example, 0 is no pain, and 10 is the worst. NPRS scores ≤ 5 correspond to mild, 6-7 to moderate, and scores ≥8 to severe pain regarding pain-related interference with functioning
Range of motion | 8 weeks
  The range of motion of the lumbosacral joint will be measured through an inclinometer for lumbar flexion (40-60 degrees), extension (20-35 degrees), and rotations (15-25 degrees) range of motion.
Posture | 8 weeks
  Leg length discrepancy (LLD) is a "direct" measurement using a tape measure that can be utilized to measure the "true" leg length from the anterior superior iliac spine (ASIS) to the medial malleolus. The "apparent" leg length is measured from the umbilicus to the medial malleolus, considered normal up to 1 cm, with mild LLD ranging from 1 to 2 cm, moderate LLD from 2 to 5 cm, and severe LLD greater than 5 cm

CONTACTS AND LOCATIONS:
Overall Officials: Faiza Amjad, PhD, Principal Investigator — Riphah international universiy
Locations (1):
- Hafiz Medical and diagnostic Center johar town Lahore, Lahore, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No